CLINICAL TRIAL: NCT04285593
Title: Efficacy of the Bulgarian Squat in the Improvement of the Asymmetries of Lower Limbs Improving the Strength in the Hamstrings and Stability of the Knees in Soccer Players. A Randomized Clinical Study.
Brief Title: Bulgarian Squat in the Improvement of Asymmetries of Lower Limbs in Soccer Players
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AJF
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Football Players
Keywords: Football; Knee; Bulgarian squat; Vertical jump; Functional movement screen; Hamstring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Each session will last 10 minutes, taking place two days a week, over a period of four weeks. The intervention will take place at the beginning of the training session.
  The players included in the experimental group will perform an exercise protocol with Bulgarian squats.
  Interventions: Other: Bulgarian squats
- Control group (No Intervention): The players included in the control group will continue with their usual warm-up routine.

INTERVENTIONS:
Other: Bulgarian squats — The intervention using Bulgarian squat exercises will consist in the application of the protocol described by Aguilera-Castells et al. The technique will be done with the footballer standing. The athlete with one foot in front and the other behind the body, arms crossed over her chest, and her upper body, will remain upright with a natural swing in the lower back during the entire exercise. The players will lower the body (eccentric phase) until the front knee flexes to 90º. Subsequently, they will return to the initial position with a full extension of the knee of the front leg (concentric phase), maintaining an erect trunk position. The front foot will be placed in a fixed position contacting the ground, and the rear foot will rest on a horizontal press bench.
  Arms: Experimental group

SUMMARY:
1541/5000 The aim of the Bulgarian squat is to improve the hamstring strength and the stability of the knees, thus reducing asymmetries in the lower limbs. It consists in achieving greater strength and stability of the lower limbs to adapt the athlete to the demands of training and competitions as safely as possible.

The main objective of the study is to assess the effectiveness of the Bulgarian squat, in the improvement of asymmetries in lower limbs; improving hamstring strength and knee stability.

Randomized, simple blind clinical study. 30 soccer players will be randomized to the study groups: experimental (Bulgarian squats) and control (non-intervention team routine). The treatment will last 4 weeks, with 2 weekly sessions of 10 minutes each. The study variables will be: lower limb strength (vertical jump with the My Jump 2 application), lower limb stability (Y ™ -Balance test) and lower limb asymmetries (Triple Hop Test, Single Hop Test for Distance and Functional Movement Screen) The normality of the sample will be calculated using the Kolmogorov -Smirnof test. The changes after each evaluation will be analyzed with the t-student test and with an ANOVA of repeated measures, the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

An improvement in the strength, stability and asymmetries of the lower limbs in soccer players is expected.

ELIGIBILITY:
Inclusion Criteria:

* Female players
* With an age range of 18 to 35 years
* Federated in the Community of Madrid
* That at the time of the study do not suffer any injury

Exclusion Criteria:

* Athletes who have not undergone surgery on the lower limbs in the last three months
* Who have not taken muscle relaxants in the last three days
* Who have not understood or have a lack of understanding about the intervention
* Have not signed the informed consent document

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline hamstring muscle strength after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done through the vertical jump Through the Appstore My Jump 2. The athlete will stand in standing position with the feet in parallel with a separation corresponding to the height of her hips. It will start with a knee flexion of 90º and with the arms along the body. You will be asked to perform a jump by bringing the lower limbs to a triple flexion (hip, knees and ankles). At the same time that it is pushed by pressing on the heels, it will take the arms in the take-off phase above its head. The load will be introduced if there is, in kg, and we will obtain the force time data (in Newton).

SECONDARY OUTCOMES:
Change from baseline stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  It will be done with the Y-Balance test. The athletes will be placed in standing position in monopodal support with a slight knee flexion in the starting platform that consists of two rear pipes that will be placed at 135º from the previous pipe with 45º between the 2 back pipes. Barefoot athletes, with the support foot behind the red line of the central starting platform, will be asked to bring the leg that is not in support to the platforms located in the anterior and posterior tubes and slide them off continuous way and without bouncing as far as you can. Six trials will be performed on each leg in each of the three directions using the highest scores for analysis. The unit of measure of this instrument is centimeters: a higher score indicates greater stability, strength and proprioception.
Change from baseline asymmetries of lower limbs after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  With the Single Hop Test for Distance we will assess the ability of the player to make a maximum monopodal jump, measuring its distance in cm. A strip of tape 15 cm wide and 6 m long perpendicular to the starting line will be placed and the athlete will rest on one leg and with her foot on the line that marks the exit by performing a maximum horizontal jump, and receiving with the same leg The arms have to be throughout the hip test, not being able to use them to improve the jump. The distance will be measured from the starting line to the back of the heel. The athlete must maintain the position after the jump for at least 3 seconds without losing balance or supporting the other leg so that the repetition is counted. In case of not fulfilling said quality criteria in the execution, the jump will be repeated after the established recovery time.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain